CLINICAL TRIAL: NCT02398357
Title: A Zelen-design Randomized Controlled Trial of the Effect of Anticoagulation After Endoscopic Therapy in Cirrhotic Patients With Portal Vein Thrombosis
Brief Title: The Effect of Anticoagulation After Endoscopic Therapy in Cirrhotic Patients With Portal Vein Thrombosis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Shiyao Chen, department of Gastroenterology, Shanghai Zhongshan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSY-LSX-2015
Record Dates: First submitted 2015-03-19; First posted 2015-03-25 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: Portal Vein Thrombosis; Liver Cirrhosis
Keywords: anticoagulation; Zelen-designed randomized controlled trial
MeSH Terms: conditions — Liver Cirrhosis | interventions — Nadroparin; Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): No anticoagulation，just routine follow-up
- Anticoagulation (Experimental): Nadroparin Calcium and Warfarin
  Interventions: Drug: Nadroparin Calcium and Warfarin

INTERVENTIONS:
Drug: Nadroparin Calcium and Warfarin — Patients will take warfarin started at a dose of 2.5mg/d and with titration of dose to maintain a target INR of 2-3,alone with Nadroparin Calcium 4100IU／d，subcutaneous, when taking endoscopy therapy .
  Arms: Anticoagulation

SUMMARY:
To determine the effect and safety of anticoagulation after endoscopic therapy in cirrhotic patients with portal vein thrombosis and to explore whether it can decrease the short-term rebleeding rate.

DETAILED DESCRIPTION:
The treatment of cirrhotic patients with PVT (portal vein thrombosis) is clearly recommended in guideline now. Several published studies has confirm the effect and safety of anticoagulation therapy in cirrhotic patients with PVT.The present studies are most observation studies with small sample size and low quality.We need more high-quality research such as randomized controlled trials. This is a Zelen-designed randomized controlled trial. Patients will randomly enter into two groups:the anticoagulation group or the control group and then we will make sure wether their are fond of the group and make decision by themselves. The recanalization rate and complications will be analyzed

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-70 years old;
* A clinical, radiological or histologic diagnosis of Liver cirrhosis and portal hypertension;
* Diagnosed of Portal vein thrombosis;
* Capable of understanding the purpose and risks of the study and informed consent to participate in the study;
* Have undergone endoscopy to prevent variceal rebleeding.

Exclusion Criteria:

* Age <18 or >70 years;
* Portal vein thrombosis diagnosed before 6 months;
* Patients with signs of acute PVT such as fever，abdominal pain or intestinal obstruction，who should be treated immediately;
* Pregnant or nursing;
* Hepatocellular carcinoma;
* Severe cardiopulmonary diseases or concomitant renal insufficiency;
* cavernous transformation of the portal vein;
* Contradictions to endoscopy;
* Contradictions to anticoagulation,such as:allergy to LMWH or warfarin, severe uncontrolled hypertension, history of hemorrhagic cerebral vascular accident, recent peptic ulcer disease, bacterial endocarditis, ulcerative colitis，sustained platelet count < 50 x103/uL);
* Taking immunosuppressive agent;
* Coagulation disorders other than the liver disease related;
* Variceal bleeding failed to control.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2015-03; Primary Completion 2017-08 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Recanalization rate of PVT | 8 weeks
  Patients will receive Doppler ultrasound before enrolled and after followed up for 8 weeks

SECONDARY OUTCOMES:
Rebleeding rate | 8 weeks
  The investigators observe the variceal rebleeding events during 8 weeks.
Incidence rate of complications | 8 weeks
  The investigators observe any severe adverse events caused by anticoagulation therapy or the progress of thrombosis.

CONTACTS AND LOCATIONS:
Overall Officials: Shiyao Chen, Professor, Study Director — Shanghai Zhongshan Hospital
Locations (1):
- Shanghai Zhongshan Hospital, Shanghai, Shanghai Municipality, China